CLINICAL TRIAL: NCT01084616
Title: The Role of Vaginal Microbiota in Symptoms of Vaginal Dryness in Postmenopausal Women
Brief Title: Vaginal Microbiota Among Postmenopausal Women
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Dr. Gregor Reid, Lawson Health Research Institute
Other Study IDs: R-09-804; 16182E (Other: Research Ethics Board)
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Last update posted 2010-12-17 (Estimated); Status verified 2010-12

CONDITIONS: Vulvovaginal Atrophy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Vaginal Dryness
- Non-vaginal dryness

SUMMARY:
It is known that vaginal bacteria have an impact upon the health status of the host, in some cases protecting against infection and in other cases causing infection, depending on the bacterial types present. This study will compare the composition of vaginal bacteria to symptoms of vaginal dryness in order to try and identify if certain bacteria might cause some of the problems associated with vaginal dryness among post-menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Between 30 and 80 years old.
* Postmenopausal = 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/ml or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.
* Prepared not to take hormone replacement therapy during 8 weeks follow-up and not taking estrogen alone or estrogen/progestin containing drug products at the time of screening.

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Reid, PhD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- Victoria Family Medical Center, London, Ontario, Canada